CLINICAL TRIAL: NCT01015079
Title: The Association Between Cervical Cancer Screening Participation and Corresponding Results and Subsequent Cancer Occurrence and Death
Brief Title: The Association Between Cervical Cancer Screening and Cancer Occurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Chi-An Chen, National Taiwan University Hospital
Other Study IDs: 200910043R
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Cervical Cancer; Cancer
Keywords: Pap smear screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Entire Taiwan women

SUMMARY:
To investigate the protective effect of cervical cancer incidence and mortality by screening attending frequency or screening pattern, and to evaluate the possible risk of developing malignancies among women with cervical lesions, inflammation or infection.

ELIGIBILITY:
The eligibility criteria in the proposal are specified in different part of analyses respectively, which are briefly listed below:

Part I:

* Include women covered by national screening program and they did not have previous cervical cancer history before the study initiate date.

Part II:

* Include women ever participated cervical cancer screening and exclude women with previous cervical cancer history before screening attending.

Part III:

* Include women without previous cervical cancer history before the follow-up initiation.

Part IV:

* Include women without previous cervical cancer history before the follow-up initiation.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The entire Taiwan women with their information obtained from several national registries.
Sampling Method: Non-Probability Sample
Enrollment: 6000000 (Estimated)
Dates: Start 2009-11

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Taiwan Cervical Cancer Screening Task Force, Taipei, Taiwan

REFERENCES:
- [Derived] Cheng WF, Chen YL, You SL, Chen CJ, Chen YC, Hsieh CY, Chen CA. Risk of gynaecological malignancies in cytologically atypical glandular cells: follow-up study of a nationwide screening population. BJOG. 2011 Jan;118(1):34-41. doi: 10.1111/j.1471-0528.2010.02769.x. Epub 2010 Nov 4. PMID 21054764